CLINICAL TRIAL: NCT02550548
Title: Incretin Action in Physiology and Diabetes
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: David D'Alessio, M.D. (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor-Investigator, David D'Alessio, M.D., Professor, Division Chief of Endocrinology, Duke University
Organization: Duke University (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: Pro00065698; R01DK101991 (NIH)
Record Dates: First submitted 2015-09-03; First posted 2015-09-15 (Estimated); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Insulin Secretion
Keywords: Incretins; GLP-1; GIP; hyperglycemic clamp; Glucagon

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- GIP infusion (Experimental): During a 240 minute hyperglycemic clamp, subjects will have (after 90 minutes of the clamp) GIP infused at 4 incremental dosages, (initial dose will be 2.0 ng/kg/min, followed by 4.0, 8.0, and 16.0 ng/kg/min). Each dose will be infused continuously for 30 minutes, followed immediately by the next higher dose. The total time of this procedure is 240 minutes.
  Interventions: Drug: GIP infusion
- GLP-1 infusion (Experimental): During a 240 minute hyperglycemic clamp, subjects will have (after 90 minutes of the clamp) GLP-1 infused at 4 incremental dosages, (initial dose will be 1.0 ng/kg/min, followed by 2.0, 3.0, and 4.0 ng/kg/min). Each dose will be infused continuously for 30 minutes, followed immediately by the next higher dose. The total time of this procedure is 240 minutes.
  Interventions: Drug: GLP-1 infusion
- GIP + GLP-1 infusion (Experimental): During a 240 minute hyperglycemic clamp, subjects will have (after 90 minutes of the clamp) GIP + GLP-1 infused simultaneously at 4 incremental dosages (doses will be half the amounts described above). These doses will be infused continuously for 30 minutes, followed immediately by the next higher doses. The total time of this procedure is 240 minutes.
  Interventions: Drug: GIP infusion; Drug: GLP-1 infusion
- GIP + Ex-9 infusion (Experimental): During a 240 minute hyperglycemic clamp, subjects will have (after 90 minutes of the clamp) GIP infused at 4 incremental dosages (as described above) with Ex-9 infused at a steady dose of 2.5 mcg/kg/min starting 90 minutes before the GIP infusion and maintained throughout the clamp experiment. The total time of this procedure is 240 minutes.
  Interventions: Drug: GIP infusion; Drug: Ex-9 infusion

INTERVENTIONS:
Drug: GIP infusion — after establishing a hyperglycemic clamp (target: 125 mg/dL) GIP will be infused
  Arms: GIP + Ex-9 infusion; GIP + GLP-1 infusion; GIP infusion
Drug: GLP-1 infusion — after establishing a hyperglycemic clamp (target: 125 mg/dL) GLP-1 will be infused
  Arms: GIP + GLP-1 infusion; GLP-1 infusion
Drug: Ex-9 infusion — Ex-9 infusion will be initiated at start of hyperglycemic clamp (target: 125 mg/dL)
  Arms: GIP + Ex-9 infusion

SUMMARY:
This project is designed to advance understanding of the incretin effect in health and disease. This system of gut-islet linkage is essential for normal glucose tolerance, impaired in T2DM, and amenable to therapeutic intervention. However, there are important gaps in understanding incretin function that limit application of this system; this project will address several of these. A secondary, but critical aspect of this research is focus on inter-individual variation in the physiology of the incretin system. This is a novel direction for research in this field and is critical to advancing the concept of individualized medical care in diabetes by establishing whether there is a physiologic basis for predicting the existence of responders and non-responders to incretin therapies.

Currently, we have described only Aim 1 from this grant in this protocol registration. While Aim 2 and 3 are described in the grant, Aim 1 will be conducted first and the results from this Aim and / or the publication of other results in the field may affect the approach to Aims 2 and 3.

ELIGIBILITY:
Inclusion Criteria:

* healthy adult volunteers
* fasting plasma glucose value ≤ 95 mg/dL, measured at screening visit
* HbA1c ≤ 5.9%, measured at screening visit

Exclusion Criteria:

* history of diabetes diagnosis, including gestational diabetes
* presence of Type II diabetes mellitus among any first degree family members
* rheumatoid arthritis
* inflammatory bowel disease
* unstable angina or uncompensated heart failure
* pulmonary disorders including COPD and asthma
* malabsorptive GI disease, such as celiac disease, or gastric bypass
* significant hepatic disease
* renal insufficiency (eGFR < 60 mL/kg/min)
* anemia (hematocrit < 34%) as measured at screening visit
* pregnancy
* uncontrolled hypertension
* consumption of daily medications that alter glucose metabolism or GI function (glucocorticoids, psychotropics, narcotics, metoclopramide)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2016-04-21 (Actual); Primary Completion 2021-04-16 (Actual); Study Completion 2021-04-16 (Actual)

PRIMARY OUTCOMES:
Beta cell sensitivity | 30 minute infusion periods
  Beta-cell sensitivity for each incretin will equal the slope of the insulin secretion rate divided by the specific incretin level (GLP-1 or GIP)

CONTACTS AND LOCATIONS:
Locations (1):
- Duke Center for Living, Durham, North Carolina, United States